CLINICAL TRIAL: NCT04423666
Title: Findings of a Health-coached Technology Based Walking Program in Unpaid Caregivers of Persons With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BostonCollege
Record Dates: First submitted 2020-05-28; First posted 2020-06-09 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Dementia
Keywords: caregiver; dementia; wellbeing; stress
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Convenience sample, randomized, intervention, pre-post design
Who Masked: Participant
Masking Description: Participants were randomly assigned through a toss of a coin to either the intervention or control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Will receive:
  1. education
  2. a wireless pedometer with set up
  3. nurse coaching via text message, email or telephone based on participant preference and at frequency determined by the participant
  Interventions: Behavioral: Walking using a wireless pedometer
- Control (Experimental): Will receive:
  1. education
  2. a wireless pedometer with set up
  Interventions: Behavioral: Walking using a wireless pedometer

INTERVENTIONS:
Behavioral: Walking using a wireless pedometer — See arm/group

SUMMARY:
This study aims to:

1. Establish the feasibility of a health-coached (HC) walking program utilizing motivational interviewing (MI) and wireless pedometers in family caregivers of persons with dementia.
2. Examine preliminary outcomes of a HC walking program utilizing MI with wireless pedometers on family caregiver's perception of wellbeing, stress, and activity level.
3. Explore caregivers' acceptability and experience of participating in a HC walking program utilizing MI with wireless pedometers and to explore additional person centered approaches.

DETAILED DESCRIPTION:
This comparative study will use a two group repeated measure design and mixed methods approach including well-validated questionnaires and qualitative descriptive methodology. Qualitative inquiry will provide data about the overall experience of caregivers in the intervention arm as well as inform web-based, person centered approaches as suggested by caregivers that will be used to inform future work on person-centered self-care strategies, aimed at improving caregiver health. Eligibility Criteria: having approval from the primary care provider to initiate a walking program, being a caregiver of a person with dementia, being greater than 18 years of age and having access to a computer or smartphone. "The "RSVP [research volunteer program] for Health," a registry comprised of individuals interested in receiving information on research studies conducted at Massachusetts General Hospital (MGH), will be utilized for recruitment. If a person states they are interested, they will be called to set up a screening visit to determine study eligibility at which time they will be given the IRB consent to review and a baseline visit will be set up.

At the baseline visit, the consent will be reviewed by the Principal Investigator (PI) and signed by participants meeting eligibility criteria. A member of the study team will obtain demographic and caregiver health characteristics and complete study questionnaires. After baseline measures are obtained, the study team will: 1) provide all participants with education about the CDC physical activity recommendations for adults, 2) set participants up with a wireless pedometer and 3) invite them to join a walking group on-line where they can monitor their activity as compared to others in the intervention arm. Members of the study team will then provide participants in the intervention arm with health coaching (HC) utilizing motivational interviewing (MI) weekly for 8 weeks by email, text message or telephone. The mode of delivery for the MI will be based on participant preference. The control group will be able to view the web page and monitor their activity compared to others in the control group arm, but will receive no coaching." At the end of the 8 weeks, study measures will be again be obtained in both groups. The PI will conduct semi-structured qualitative interviews with participants in the intervention arm to evaluate acceptability and acquire feedback on the intervention and ideas for other self-care strategies." Caregiver Measures Pre - Post

1. Demographic variables
2. General health characteristics
3. Well-being
4. Perceived stress
5. Mini-cog
6. Perceived Steps And post, a qualitative interview

ELIGIBILITY:
Inclusion Criteria - must have/be:

Approval from the primary care provider to initiate a walking program A caregiver of a person with dementia Greater than age 18 Access access to a computer or smartphone.

Exclusion Criteria:

Not being able to commit to an 8 week walking program

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 8 weeks
  systolic/diastolic
Pulse rate will be combined to report BMI in kg/m^2BMI | 8 weeks
  count of pulse rate for one minute
height | 8 weeks
  in meters
weight | 8 weeks
  in kg
BMI | 8 weeks
  weight and height will be combined to report BMI in kg/m^2

SECONDARY OUTCOMES:
wellbeing | 8 weeks
  self report using 7 item Warwick wellbeing where 1 is none to 5 is all of the time (more positive reponse)
Stress level | 8 weeks
  self report using 10-item Perceived Stress Scale where 1 is no stress to 4 is highest level of stress
Qualitative Descriptive | At end of 8 weeks
  interviews

CONTACTS AND LOCATIONS:
Overall Officials: Jane Flanagan, PhD, Principal Investigator — Boston College
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Pi will make available upon request the study protocol, SAP, ICF and CSR and as possible these will be shared via dissemination of the findings.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: April 2020 - indefinitely
Access Criteria: notify PI
URL: http://www.bc.edu/bc-web/schools/cson/faculty-research/faculty-directory/jane-m--flanagan.html